CLINICAL TRIAL: NCT06883955
Title: Prospective Cohort Study of the Clinical Features and Current Treatment of Primary Headache
Brief Title: Clinical Features and Current Treatment of Primary Headache
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yamei Tang, Professor and Associate Dean, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSKY-2025-081-01
Record Dates: First submitted 2025-03-05; First posted 2025-03-19 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Primary Headache
Keywords: primary headache; prospective cohort study; clinical features; current treatment
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Years
Biospecimen Retention: Samples With DNA — Freshly collect the blood and feces of patients with primary headache to detect biomarker changes, including white blood cell quantification and classification, inflammatory indicators, and fecal bacteriological examination.
  For imaging biomarker changes: Observe changes in brain structure, brain function, and metabolism.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- primary headache: Subjects who are younger than 65 years old and meet the diagnostic criteria for relevant primary headaches (such as tension-type headache, migraine, cluster headache, trigeminal autonomic cephalalgia, etc.) in the third edition of the International Classification of Headache Disorders (ICHD-3).
  Interventions: Combination Product: Disease education, pharmacological treatment, Non-pharmacological treatment

INTERVENTIONS:
Combination Product: Disease education, pharmacological treatment, Non-pharmacological treatment — Disease education: Provide patients with education on knowledge related to primary headache, including the causes, pathogenesis, symptoms, treatment methods, and preventive measures of headache, etc., to help patients better understand their own diseases and improve their self-management ability.
  Non-pharmacological treatment: Although specific non-pharmacological treatment methods are not elaborated in detail in the research protocol, they may include psychotherapy, physical therapy, etc. For example, biofeedback therapy, relaxation training, transcranial magnetic stimulation, etc. These can all be recorded as possible intervention measures.
  Pharmacological treatment: Record the medications used for the treatment of acute episodes and preventive treatment by patients during the research process, including the types of medications, dosages, frequency of use, etc. For instance, non-steroidal anti-inflammatory drugs and triptan drugs used during acute episodes, and β-blockers.

SUMMARY:
This study is a prospective, observational cohort study. The plan of this study is to consecutively enroll 2,000 primary headache patients who meet the inclusion criteria from the neurology outpatient department and inpatient department of Sun Yat-sen Memorial Hospital, Sun Yat-sen University. Basic clinical data registration, various scale evaluations, cranial imaging examinations, and collection of blood and fecal biological samples will be completed. During the 10-year follow-up plan, systematic clinical evaluations of the disease severity, diagnosis and treatment, living ability and health status of patients will be carried out regularly every 6 - 12 months. Imaging and other functional evaluations will be conducted when necessary. Data collection includes:

Demographic data (including age, gender, education, ethnicity, marital status, occupation, etc.); General clinical data (past medical history, medication history, personal history, menstrual and childbearing history, family history, etc.); Clinical data of primary headache: headache frequency, duration, severity (Numeric Rating Scale for pain, NRS), headache-related medication use, drug efficacy and side effects; Scale evaluations: MIDAS, HIT-6, BPI, MSQ, ADL, CDR, PGIC, CGIC, PHQ-4, mTOQ-4, ASC-12, MIBS-4, HARDSHIP, WHO-QOL BREF, HAMD, HAMA, TNQ; Records of neurological imaging examinations, blood sample and fecal sample collection.

DETAILED DESCRIPTION:
Background Headache is one of the most common diseases in the nervous system. Approximately 52% of adults worldwide suffer from primary headache. The third edition of the International Classification of Headache Disorders in 2018 classified primary headache into migraine, tension-type headache, trigeminal autonomic cephalalgia, and other primary headaches. Although primary headache has no obvious organic lesions, it can lead to transient or permanent central nervous system dysfunction, affecting people's daily life and work, and imposing a huge economic burden on society. This study intends to establish a prospective cohort of patients with primary headache, observe the relevant risk factors, clinical treatment efficacy, and prognosis of patients with primary headache, and explore the relevant clinical factors and biomarkers for a favorable prognosis. During the 10-year follow-up plan, systematic clinical evaluations will be regularly carried out on the disease severity, diagnosis and treatment status, living ability, and health status of patients. When necessary, blood and fecal samples will be collected and imaging evaluations will be conducted to complete the construction of a clinical diagnosis and treatment information database for patients with primary headache, and analyze the clinical factors related to the prognosis.

Research Objectives To observe the risk factors, clinical characteristics, treatment regimens and their efficacy, and prognosis of patients with primary headache, and to explore the relevant clinical factors and biomarkers for a favorable prognosis.

Research Design This study adopts a single-center, prospective cohort design.

Baseline Assessment Demographic data (including: age, gender, education level, ethnicity, marital status, occupation, etc.); General clinical data (past medical history, medication history, personal history, menstrual, marital and childbearing history, and family history, etc.); Clinical data of primary headache: headache frequency, duration, severity (Numerical Rating Scale for Pain, NRS), past headache-related medication use, medication efficacy and side effects; Scale Evaluation: MIDAS, HIT-6, BPI, MSQ, ADL, CDR, PGIC, CGIC, PHQ-4, mTOQ-4, ASC-12, MIBS-4, HARDSHIP, WHO-QOL BREF, HAMD, HAMA, TNQ; Biochemical Indicators: White blood cell count and classification, inflammatory indicators in the blood; fecal bacteriological examination; Changes in Imaging Biomarkers: Changes in brain structure, brain function, and metabolism.

Follow-up Study

Within 6 months after enrollment, follow-up assessments will be conducted every 1-3 months; from half a year to 10 years after enrollment, follow-up assessments will be conducted every 6-12 months (the assessment methods include in-person interviews, telephone follow-ups, and online follow-ups). The following data will be collected:

Clinical data of primary headache: headache frequency, duration, severity (Numerical Rating Scale for Pain, NRS), the use of headache-related medications (types, dosages, efficacy, and side effects); Scale Evaluation: MIDAS, HIT-6, BPI, MSQ, ADL, CDR, PGIC, CGIC, PHQ-4, mTOQ-4, ASC-12, MIBS-4, HARDSHIP, WHO-QOL BREF, HAMD, HAMA, TNQ; Blood and fecal tests and cranial imaging examinations (when clinically necessary and with the patient's/family member's consent and cooperation).

ELIGIBILITY:
Inclusion Criteria:

1. Age is less than 65 years old.
2. Meets the diagnostic criteria for relevant primary headaches (such as tension-type headache, migraine, cluster headache, trigeminal autonomic cephalalgia, etc.) in the third edition of the International Classification of Headache Disorders (ICHD - 3).
3. Is willing and able to participate throughout the entire study period and sign the informed consent form.
4. Has the ability to complete the "Headache Diary" independently or with the help of a guardian.

Exclusion Criteria:

1. Secondary headache
2. High - risk populations, such as those with severe heart disease, impaired liver and kidney function, malignant tumors, etc.
3. Patients with mental illness, cognitive impairment, or those who are unable to cooperate with the research requirements
4. History of intracranial lesions or other nervous system diseases (including stroke, epilepsy, etc.)

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary headache is a common neurological disease worldwide, with a prevalence rate of approximately 10% - 20%. Its occurrence is not related to brain structural damage, infection, metabolic abnormalities, or other diseases, but is directly caused by the abnormal function of the central or peripheral nervous system. According to the ICHD-3, primary headache mainly includes migraine, tension - type headache, and cluster headache etc. The attack frequency, duration, and severity of primary headache show a high degree of heterogeneity. Primary headache is highly comorbid with anxiety, depression, and sleep disorders. The quality of life of patients with chronic primary headache significantly declines, and the work absenteeism rate and economic burden increase. Analgesic drugs are mainly used in the acute phase. Preventive treatment is applicable to patients with frequent or chronic attacks, and non-pharmacological interventions are also effective strategies.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-03-08 (Estimated); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
The number of headache days per month. | 10 years
  The number of headache days per month: This indicator is used to count the actual number of days each research subject experiences headache symptoms within each month. Through the recording and analysis of the number of headache days per month, it can directly reflect the frequency of headache attacks, helping researchers understand the duration of the interference of primary headache with the daily life of patients, and further evaluate the severity and development trend of the disease.
Changes in scores of headache assessment scales: NRS. | 10 years
  NRS (The Numerical Rating Scale for Pain) is a commonly used simple pain measurement tool. Patients select a value within the numerical range from 0 (representing no pain) to 10 (representing the most severe pain) according to the degree of pain they feel, to quantify the intensity of pain.
Changes in scores of headache assessment scales: HIT-6. | 10 years
  The HIT - 6 scale (the Headache Impact Test - 6) is mainly used to evaluate the impact of headache on various aspects of patients' lives, such as daily activities, social interaction, work, etc.

SECONDARY OUTCOMES:
The number of days of emergency medication use per month. | 10 years
The types of preventive medications and the number of days of use per month. | 10 years
Changes in scale scores at MIDAS. | 10 years
  Changes in scale scores at Migraine Disability Assessment Scale (MIDAS)
Changes in scale scores at BPI. | 10 years
  Changes in scale scores at Brief Pain Inventory (BPI).
Changes in scale scores at MSQ. | 10 years
  Changes in scale scores at Migraine Specific Quality of Life Questionnaire (MSQ).
Changes in scale scores at PGIC and CGIC. | 10 years
  Changes in scale scores at Patient Global Impression of Change (PGIC) and Clinician Global Impression of Change (CGIC).
Changes in scale scores at HAMD and HAMA. | 10 years
  Changes in scale scores at Hamilton Depression Rating Scale (HAMD) and Hamilton Anxiety Rating Scale (HAMA).
Changes in scale scores at WHO - QOLBREF. | 10 years
  Changes in scale scores at World Health Organization Quality of Life - BREF (WHO - QOL BREF).
Changes in scale scores at HARDSHIP. | 10 years
  Changes in scale scores at Headache - Related Disability Scale (HARDSHIP).
Concentration of White Blood Cell Count and Subtypes in Peripheral Blood. | 10 years
  Absolute counts (×10^9/L) and percentage (%) of neutrophils, lymphocytes, monocytes, eosinophils, and basophils.
Change in serum inflammatory cytokine levels. | 10 years
  Concentration of pro-inflammatory cytokines (IL-6, TNF-α, CRP) in serum measured by chemiluminescence immunoassay.
Diversity and Abundance of Fecal Microbiota. | 10 years
  Shannon index (unitless), Firmicutes/Bacteroidetes ratio (%).
Change in gray matter volume. | 10 years
  Regional gray matter volume in pain-processing areas (insula, thalamus, anterior cingulate cortex) quantified by voxel-based morphometry (VBM) on 3T MRI.
Change in resting-state functional connectivity. | 10 years
  Functional connectivity strength within the default mode network (DMN) measured by fMRI BOLD signal.
Change in brain metabolic profile. | 10 years
  Concentration ratio of N-acetylaspartate (NAA) to creatine (Cr) in the thalamus measured by proton magnetic resonance spectroscopy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stovner LJ, Hagen K, Linde M, Steiner TJ. The global prevalence of headache: an update, with analysis of the influences of methodological factors on prevalence estimates. J Headache Pain. 2022 Apr 12;23(1):34. doi: 10.1186/s10194-022-01402-2. PMID 35410119
- [Background] Steiner TJ, Stovner LJ, Jensen R, Uluduz D, Katsarava Z; Lifting The Burden: the Global Campaign against Headache. Migraine remains second among the world's causes of disability, and first among young women: findings from GBD2019. J Headache Pain. 2020 Dec 2;21(1):137. doi: 10.1186/s10194-020-01208-0. No abstract available. PMID 33267788